CLINICAL TRIAL: NCT03645434
Title: A Phase IIa, Randomised, Multi-centre, Double-blind, Placebo and Active-controlled, 3 Periods, Crossover Study to Investigate the Efficacy, Pharmacokinetics, Safety and Tolerability of Inhaled AZD8871 Administered Once Daily for 2 Weeks in Patients With Moderate to Severe COPD
Brief Title: A Single Inhalation Dose Study to Assess Efficacy, Pharmacokinetics (PK), Safety and Tolerability of AZD8871 in Patients With Long-term Lung Diseases.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D6640C00006
Record Dates: First submitted 2018-08-09; First posted 2018-08-24 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Moderate to severe COPD; Muscarinic receptor antagonist; β2 adrenoceptor agonist (MABA); Long-acting muscarinic antagonist (LAMA); Long-acting β2-agonist (LABA); Inhaled long-acting bronchodilator; Small airways disease (obstructive bronchiolitis); Parenchymal destruction (emphysema),
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — AZD-8871; vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This study will be performed in a double-blind manner. Each investigational product (IP) and its placebo will be supplied in identical packaging to enable double-blind conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment sequence A (Experimental): Randomized patients will receive multiple oral dose of inhalation powder via DPI as follow:
  Treatment period 1: AZD8871 600 µg and Anoro® Ellipta® matching placebo.
  Treatment period 2: AZD8871 matching placebo and Anoro® Ellipta® 55 μg / 22 μg.
  Treatment period 3: Matching placebo of AZD8871 and Anoro® Ellipta®
  Interventions: Drug: AZD8871; Drug: Anoro® Ellipta®
- Treatment sequence B (Experimental): Randomized patients will receive multiple oral dose of inhalation powder via DPI as follows:
  Treatment period 1: AZD8871 600 µg and Anoro® Ellipta® matching placebo.
  Treatment period 2: Matching placebo of AZD8871 and Anoro® Ellipta®
  Treatment period 3: AZD8871 matching placebo and Anoro® Ellipta® 55 μg / 22 μg.
  Interventions: Drug: AZD8871; Drug: Anoro® Ellipta®
- Treatment sequence C (Experimental): Randomized patients will receive multiple oral dose of inhalation powder via DPI as follows:
  Treatment period 1: AZD8871 matching placebo and Anoro® Ellipta® 55 μg / 22 μg.
  Treatment period 2: AZD8871 600 µg and Anoro® Ellipta® matching placebo.
  Treatment period 3: Matching placebo of AZD8871 and Anoro® Ellipta®
  Interventions: Drug: AZD8871; Drug: Anoro® Ellipta®
- Treatment sequence D (Experimental): Randomized patients will receive multiple oral dose of inhalation powder via DPI as follow:
  Treatment period 1: AZD8871 matching placebo and Anoro® Ellipta® 55 μg / 22 μg.
  Treatment period 2: Matching placebo of AZD8871 and Anoro® Ellipta®
  Treatment period 3: AZD8871 600 µg and Anoro® Ellipta® matching placebo.
  Interventions: Drug: AZD8871; Drug: Anoro® Ellipta®
- Treatment sequence E (Experimental): Randomized patients will receive multiple oral dose of inhalation powder via DPI as follow:
  Treatment period 1: Matching placebo of AZD8871 and Anoro® Ellipta®
  Treatment period 2: AZD8871 600 µg and Anoro® Ellipta® matching placebo.
  Treatment period 3: AZD8871 matching placebo and Anoro® Ellipta® 55 μg / 22 μg.
  Interventions: Drug: AZD8871; Drug: Anoro® Ellipta®
- Treatment sequence F (Experimental): Randomized patients will receive multiple oral dose of inhalation powder via DPI as follow:
  Treatment period 1: Matching placebo of AZD8871 and Anoro® Ellipta®
  Treatment period 2: AZD8871 matching placebo and Anoro® Ellipta® 55 μg / 22 μg.
  Treatment period 3: AZD8871 600 µg and Anoro® Ellipta® matching placebo.
  Interventions: Drug: AZD8871; Drug: Anoro® Ellipta®

INTERVENTIONS:
Drug: AZD8871 — Randomized patients will receive 14 repeated daily doses of AZD8871 600 µg inhalation powder via DPI.
Drug: Anoro® Ellipta® — Randomized patients will receive 14 repeated daily doses of Anoro® Ellipta® (55 µg/22 µg) inhalation powder via DPI.
  Other Names: Anoro® - Umeclidinium/Vilanterol; Ellipta® - Device

SUMMARY:
This study will evaluate the efficacy and safety data of AZD8871 in patients with moderate to severe chronic obstructive pulmonary disease (COPD). This study will determine the 24-hour efficacy (lung function) profile of AZD8871 600 μg relative to placebo dry powder inhaler (DPI) based on trough forced expiratory volume in 1 second (FEV1) following repeated dosing (2 weeks). Anoro® Ellipta® (umeclidinium/vilanterol) once daily is included as an active control. This study aims at providing a novel approach to the treatment of COPD with greater efficacy than single-mechanism bronchodilators, equivalent to long-acting muscarinic antagonist (LAMA) and long-acting β2-agonist (LABA) administered as free- or fixed-dose combination therapies, with an equivalent or superior safety and tolerability profile.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo and active-controlled crossover study will be conducted at 5 sites in Germany and the United Kingdom (UK). Approximately 180 patients will be screened in order to randomize 72 patients into the study. Based on previous studies estimate, it is anticipated that 54 patients will be evaluable (study completers) assuming an approximate 25% dropout rate. A subset of 36 patients, who will have specifically consented for pharmacokinetics (PK), will undergo PK assessments. The study will consist of -

* A Screening period: Will last up to 28 days and consists of 2 Screening visits (Visit 1 and Visit 2) and a run-in period (between a minimum of 14 and a maximum of 28 days; from Visit 2 to Visit 3).
* Three treatment periods (Visit 3; 14 days each; each separated by a wash-out period of 42 to 49 days) and
* A Follow-up Visit: 42 days (up to 49 days) after last investigational product (IP) administration.

Patients will be requested to stop their usual COPD therapy after signing the informed consent form (ICF) at Visit 1 and will be maintained on a mono-component inhaled corticosteroid (ICS) therapy, if required. Patients that were taking any LAMA will be maintained with ipratropium (34 µg × 2 puffs 4 times per day) between Visit 1 and Visit 2. In addition, salbutamol 100 µg will be provided as rescue medication during the study as needed (rescue medication has to be discontinued 6 hours before any pulmonary function test). Visit 1 and Visit 2 could be performed on the same day if no wash-out of prior medication is required and the patient visits the site in fasting condition. In case any wash-out of prior medication is required, then Visit 2 will be performed after the wash-out is complete. If reversibility criteria and forced expiratory volume in 1 second (FEV1) predicted values are fulfilled according to inclusion criteria, the patient will be started on run-in period to assess clinical stability. If reversibility criteria or FEV1 predicted values are not met, pulmonary function tests could be rescheduled at the latest, up to Day 14. During the run in period, all patients will receive ipratropium 34 µg × 2 puffs 4 times per day (must be discontinued 8 hours prior to previous any pulmonary function test). A paper diary will be used to collect adverse events (AEs) and concomitant medication during run-in and wash-out periods.

Eligible patients will be randomized in 1:1:1:1:1:1 ratio to 1 of 6 treatment sequences and will receive orally 1 of the following 3 treatments sequence in the form of inhalation powder using DPI :

* AZD8871 600 µg once daily (double-blind).
* Anoro® Ellipta® (55 µg umeclidinium [UMEC]/ 22 µg vilanterol [VI]) once daily (double-blind).
* Placebo (double-blind). Study treatment administration during all the visits at the sites (Day 1, Day 2, Day 8, and Day 14 of each treatment period) will be supervised by study personnel.

During the treatment period Visits, safety and tolerability assessments and pulmonary function measurements will be taken pre-dose and up to 24 hours (Day 1) and up to 4 hours (Day 8) post-dose, respectively.

At Visits 3 to 11, a subset of 36 patients will undergo PK assessments. Blood samples will be collected pre-dose and up to 24 hours post dose.

In follow-up visit, AEs, safety laboratory, electrocardiogram (ECG), vital signs and physical examination will be assessed.

The study includes 12 visits and the entire study period is scheduled to take from a minimum of 6.5 months (182 days) to a maximum of 7.5 months (217 days) for each individual patient. The estimated study duration is 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written ICF prior to any study-specific procedures, sampling, and analyses.
2. Patient must be 40 to 85 years male and/or females of non-childbearing potential who are not pregnant/lactating at the time of signing the ICF (Screening; Visit 1).
3. Patient with an established clinical history of moderate to severe COPD for more than 1 year at Screening, according to the GOLD COPD guidelines.
4. Patient who is a current or former smoker (defined as one who has stopped smoking for at least 6 months prior to Screening) with a history of ≥10 pack-years of cigarette smoking [Number of pack-years=(number of cigarettes per day/20)* number of years smoked (eg, 1 pack-year=20 cigarettes smoked per day for 1 year)].
5. Patient with post-bronchodilator FEV1/forced vital capacity (FVC) ratio <70% based on the value reached after inhalation of salbutamol (400 µg) at Visit 2. If criterion is not met, the test can be repeated at the latest, up to Day -14.
6. Patient with post-bronchodilator FEV1 that must be ≥40% and <80% predicted normal value at Visit 2. If criterion is not met, the test can be repeated at the latest, up to Day -14.
7. Patient is willing and, in the opinion of the Investigator, able to change current COPD therapy as required by the protocol and willing to use ipratropium following the approved dosage and regimen (during run-in and wash-out periods) with or without ICS for maintenance therapy of COPD and rescue medication salbutamol (as needed) from Visit 1 to Visit 11.
8. Patient must be able to read, speak and understand local language, and be willing to remain at the study centre as required per-protocol to complete all visit assessments.
9. Body mass index (BMI) <40 kg/m2 at the time of Screening.
10. Female patients must be of non-childbearing potential defined as:

    * Permanently or surgically sterilised, including hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy.
    * Post-menopausal; aged <50 years and amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post menopausal range of the local laboratory.
    * Post-menopausal; aged ≥50 years and amenorrhoeic for 12 months or more, following cessation of all exogenous hormonal treatments.
11. Male patients should use a condom and spermicide to prevent pregnancy and drug exposure of a partner, regardless of the gender or childbearing potential of the partner from the day of the first administration of the IP until 3 months after the last administration of the IP. In addition to a condom with spermicide, a second highly effective method of contraception (oral, intravaginal or transdermal hormonal contraceptives, intrauterine device, intrauterine hormone-releasing system, or sexual abstinence until 3 months after the last administration of the IP) should be used with female partners of childbearing potential. Double barrier methods (a combination of male condom with either a cap, diaphragm or sponge with spermicide) are not considered to be highly effective methods of contraception. Male patients with a pregnant partner should use a condom and spermicide.

Exclusion Criteria:

1. Patient has significant diseases other than COPD, (ie, clinically relevant disease or condition or an abnormality in prior ECGs, medical history or physical examinations) which, in the opinion of the Investigator, may put the patient at risk because of participation in the study or may influence either the results of the study or the patient's ability to participate in the study.
2. Patient has alpha-1 antitrypsin deficiency as the cause of COPD.
3. Patient has other active pulmonary disease such as predominant asthma, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, idiopathic interstitial pulmonary fibrosis, primary pulmonary hypertension, or uncontrolled sleep apnoea. Allergic rhinitis is not exclusionary.
4. Lung surgery for volume reduction or lung transplantation: Patient has undergone lung volume reduction surgery, lobectomy, or bronchoscopic lung volume reduction (endobronchial blockers, airway bypass, endobronchial valves, thermal vapour ablation, biological sealants, massive pulmonary embolism and airway implants) within 1 year of Screening (Visit 1).
5. Patient is using nocturnal positive pressure (eg, continuous positive airway pressure or bi level positive airway pressure). Patient is using any non-invasive positive pressure ventilation device. Note: A patient using continuous positive airway pressure or bi level positive airway pressure for Sleep Apnoea Syndrome is allowed in the study.
6. Patient who had 2 or more exacerbations of COPD (moderate or severe in intensity) within the last year prior to Screening (see Section 7.1 for definition of exacerbation of COPD).
7. Patient has been hospitalised due to poorly controlled COPD within 3 months of the Screening period.
8. Patient has acute worsening of COPD that requires treatment with corticosteroids or antibiotics in the 6 week interval prior to or during the Screening period.
9. Patient has had lower respiratory tract infection(s) that required antibiotics within 6 weeks prior to the Screening period.
10. Patient has significant cardiovascular disease that may be vulnerable to cardiovascular instability. Note: Some examples of clinically significant cardiovascular conditions are:

    * Myocardial infarction within the 6 months prior to Screening Visit (Visit 1).
    * Unstable angina or unstable arrhythmia which has required changes in the pharmacological therapy or other intervention within 12 months prior to Screening (Visit 1), or newly diagnosed arrhythmia within the previous 3 months prior to Screening (Visit 1).
    * Second degree atrio-ventricular block.
    * Use of pacemaker.
    * Hospitalisation within 12 months prior to Screening (Visit 1) for heart failure functional classes III (marked limitation of activity and only comfortable at rest) and IV per the "New York Heart Association".
11. Patient with a QT interval corrected using Fridericia's formula (QTcF) value >450 ms for male and >470 ms for female or an ECG that is not suitable for QT measurements (eg, poorly defined termination of the T wave).
12. Patient with a heart rate <50 or >120 beats per minute (bpm).
13. Patient has clinically significant uncontrolled hypertension (>180 mmHg) as assessed by the Investigator.
14. Patient has seizures or a history of seizures requiring anticonvulsants within 12 months prior to Screening.
15. Patient is taking selective serotonin reuptake inhibitors or serotonin-norepinephrine reuptake inhibitors whose dose has not been stable for at least 4 weeks prior to Screening, or exceeds the maximum recommended dose.
16. Patient has a symptomatic bladder neck obstruction, acute urinary retention or symptomatic non-stable prostate hypertrophy.
17. Any laboratory abnormality or suspicion of any clinically relevant disease or disorder (on history or examination), including uncontrolled diabetes or hypokalaemia (serum potassium <3.5 mmol/L), which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study, or any other safety concerns in the opinion of the Investigator. Note: Potassium replacement and re-test is allowed once if serum potassium concentration was <3.5 mmol/L at Screening or prior to randomisation.
18. Patient has known human immunodeficiency virus (HIV) infection or chronic hepatitis B or C infection.
19. History of malignancy of any organ system, treated or untreated within the past 5 years, with the exception of localised basal cell carcinoma of the skin.
20. Patient has known narrow-angle glaucoma.
21. Patient has a history of drug of abuse within the past 2 years or consuming more than 14 (female patients) or 21 (male patients) units of alcohol a week, or shows positive for drugs of abuse and alcohol tests at Screening and prior to randomisation.

    Note: If a patient tests positive to any drugs of abuse tests, which cannot be explained by use of prescription medication, he/she will be excluded from the study. Unit=1 glass of wine (125 mL)=1 measure of spirits=½ pint of beer.
22. Patient has a history of hypersensitivity (including paradoxical bronchospasm) to β2-agonists, muscarinic anticholinergics or lactose/milk protein. Lactose intolerance is not an exclusion criterion.
23. Patient has received a live attenuated vaccination within 30 days prior to Screening.

    Note: Inactivated influenza vaccination, pneumococcal vaccination, or any other inactivated vaccine is acceptable provided it is not administered within 7 days prior to Screening or randomisation (Visit 3).
24. Patient who, in the opinion of the Investigator, is unable to abstain from protocol-defined prohibited medications during the study.
25. Patient was treated with an investigational drug or device in another clinical trial within the last 30 days or 5 half-lives (whichever is longer) prior to Screening.

    Note: Patient participation in observational studies (ie, studies that do not require change to medication or an additional intervention) is not exclusionary.
26. Previous participation or prior screen failure in the present study.
27. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
28. Patient has changed their smoking status (ie, restarted or stopped smoking) or initiation of a smoking cessation program within 6 weeks of Screening.
29. Patient has participated in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Screening or who will enter the acute phase of a pulmonary rehabilitation program during the study. A patient in the maintenance phase of a pulmonary rehabilitation program is not to be excluded.
30. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements. Inability to comply with requirements includes having an e-Diary completion rate of <70% during the run-in period.
31. Patient who have donated or lost >500 mL of blood and/or plasma within the previous 3 months prior to Screening.
32. Vulnerable patients (who has been placed in an institution due to a regulatory or court order).

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (3):
  - Research Site, Berlin
  - Research Site, Grosshansdof
  - Research Site, Wiesbaden
- United Kingdom (2):
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Singh D, Beier J, Astbury C, Belvisi MG, Da Silva CA, Jauhiainen A, Jimenez E, Lei A, Necander S, Smith JA, Wahlby Hamren U, Xin W, Psallidas I. The novel bronchodilator navafenterol: a phase 2a, multicentre, randomised, double-blind, placebo-controlled crossover trial in COPD. Eur Respir J. 2022 Apr 7;59(4):2100972. doi: 10.1183/13993003.00972-2021. Print 2022 Apr. PMID 34503985
- See also: Redacted SAP. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6640C00006&attachmentIdentifier=1e159c5a-28c2-4e30-ab31-be619599cfe8&fileName=D6640C00006_PXL_240583_Final_Draft_redacted_SAP_10June2020.pdf&versionIdentifier=
- See also: Redacted CSP. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6640C00006&attachmentIdentifier=cb3ce046-d8ba-426c-98dd-a898051d2456&fileName=D6640C00006_PXL_240583_Final_Draft_redacted_CSP_10June2020.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who met all the inclusion and none of the exclusion criteria were enrolled at 3 sites in Germany and 2 sites in the United Kingdom (UK).
Pre-assignment Details: Subjects attended Screening Visit within a 14 to 28-days Screening Period, before receiving their first dose of AZD8871. All subjects underwent inclusion exclusion criteria assessment and all eligible subjects signed the informed consent before undergoing any study related procedures.
Groups:
- Treatment Sequence A: Randomized subjects received 14 repeated daily oral doses of inhalation powder via DPI as follows:
  Treatment period 1: AZD8871 600 μg and Anoro® Ellipta® matching placebo. Treatment period 2: AZD8871 matching placebo and Anoro® Ellipta® 55 μg / 22 μg. Treatment period 3: Matching placebo of AZD8871 and Anoro® Ellipta®.
- Treatment Sequence B: Randomized subjects received 14 repeated daily oral doses of inhalation powder via DPI as follows:
  Treatment period 1: AZD8871 600 μg and Anoro® Ellipta® matching placebo. Treatment period 2: Matching placebo of AZD8871 and Anoro® Ellipta®. Treatment period 3: AZD8871 matching placebo and Anoro® Ellipta® 55 μg / 22 μg.
- Treatment Sequence C: Randomized subjects received 14 repeated daily oral doses of inhalation powder via DPI as follows:
  Treatment period 1: AZD8871 matching placebo and Anoro® Ellipta® 55 μg / 22 μg.
  Treatment period 2: AZD8871 600 μg and Anoro® Ellipta® matching placebo. Treatment period 3: Matching placebo of AZD8871 and Anoro® Ellipta®.
- Treament Sequence D: Randomized subjects received 14 repeated daily oral doses of inhalation powder via DPI as follows:
  Treatment period 1: AZD8871 matching placebo and Anoro® Ellipta® 55 μg / 22 μg.
  Treatment period 2: Matching placebo of AZD8871 and Anoro® Ellipta®. Treatment period 3: AZD8871 600 μg and Anoro® Ellipta® matching placebo.
- Treatment Sequence E: Randomized subjects received 14 repeated daily oral doses of inhalation powder via DPI as follows:
  Treatment period 1: Matching placebo of AZD8871 and Anoro® Ellipta®. Treatment period 2: AZD8871 600 μg and Anoro® Ellipta® matching placebo. Treatment period 3: AZD8871 matching placebo and Anoro® Ellipta® 55 μg / 22 μg.
- Treatment Sequence F: Randomized subjects received 14 repeated daily oral doses of inhalation powder via DPI as follows:
  Treatment period 1: Matching placebo of AZD8871 and Anoro® Ellipta®. Treatment period 2: AZD8871 matching placebo and Anoro® Ellipta® 55 μg / 22 μg. Treatment period 3: AZD8871 600 μg and Anoro® Ellipta® matching placebo.
Period: Period 1
Arm/Group | Treatment Sequence A | Treatment Sequence B | Treatment Sequence C | Treament Sequence D | Treatment Sequence E | Treatment Sequence F
Started | 12 | 13 | 13 | 11 | 12 | 12
Completed | 12 | 13 | 13 | 10 | 11 | 12
Not Completed | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — COPD exacerbation | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Treatment Sequence A | Treatment Sequence B | Treatment Sequence C | Treament Sequence D | Treatment Sequence E | Treatment Sequence F
Started | 10 (2 subject discontinued as they did not meet stability or FEV1 variability.) | 13 | 13 | 10 | 11 | 11 (1 subject completed Period 1 but not allowed to enter Period 2 due to physician decision.)
Completed | 10 | 13 | 13 | 10 | 11 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Treatment Sequence A | Treatment Sequence B | Treatment Sequence C | Treament Sequence D | Treatment Sequence E | Treatment Sequence F
Started | 10 | 13 | 11 (2 subjects discontinued as they did not meet FEV1 stability criteria or pfts variability criteria.) | 10 | 11 | 11
Completed | 10 | 13 | 11 | 10 | 11 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Subjects received AZD8871 inhalation powder 600 μg, 1 inhalation per day; umeclidinium 55 μg / vilanterol 22 μg. as oral inhalation once per day; Placebo to AZD8871 via oral inhalation, 1 inhalation per day.
Arm/Group | All Participants
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.0 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 73
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough FEV1 at Day 15
Description: To evaluate the efficacy of inhaled AZD8871 600 μg in patients with moderate to severe chronic obstructive pulmonary disease (COPD).
Time Frame: Day 15
Population: The full analysis set (FAS): All participants randomised and receiving study treatment, irrespective of their protocol adherence and continued participation in the study.
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- AZD8871: Subjects received AZD8871 (as saccharinate) inhalation powder 600 μg, orally 1 inhalation per day in treatment period 1 under sequences A and B; treatment period 2 under sequences C and E; and treatment period 3 under sequences D and F.
- Anoro® Ellipta®: Subjects received Anoro® Ellipta® (umeclidinium / vilanterol) 55 μg / 22 μg orally 1 inhalation per day in treatment period 1 under sequences C and D; treatment period 2 under sequences A and F; and treatment period 3 under sequences B and E.
- Placebo: Placebo to AZD8871 and Anoro® Ellipta® orally 1 inhalation per day in treatment periods 1, 2 and 3 under all sequences A, B; C, D, E and F.
Arm/Group | AZD8871 | Anoro® Ellipta® | Placebo
Number analyzed (Participants) | 70 | 69 | 68
Liters | 0.1904 (0.2052) | 0.2260 (0.2275) | -0.0222 (0.1404)
Statistical Analysis 1: Comparison: AZD8871 vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.202, 95% CI 2-sided [0.151 to 0.253]

2. Secondary Outcome: FEV1 AUC(0-4)/4h (Area Under the Curve for the Change in FEV1 From Baseline to 4h, Normalised by the Time Window)
Description: To evaluate the efficacy of inhaled AZD8871 600 μg in patients with moderate to severe COPD
Time Frame: At Day 1, Day 8, and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | AZD8871 | Anoro® Ellipta® | Placebo
Number analyzed (Participants) | 70 | 69 | 68
Liters
  Day 1: number analyzed (Participants) | 69 | 69 | 67
  Day 1 | 0.3604 (0.1753) | 0.2912 (0.1677) | 0.0430 (0.0783)
  Day 8 | 0.4296 (0.2197) | 0.3796 (0.2133) | 0.0808 (0.2117)
  Day 14: number analyzed (Participants) | 70 | 68 | 67
  Day 14 | 0.4060 (0.2448) | 0.3358 (0.2011) | 0.0209 (0.1210)

3. Secondary Outcome: FEV1 AUC(0-8)/8h (Area Under the Curve for the Change in FEV1 From Baseline to 8h, Normalised by the Time Window)
Description: To evaluate the efficacy of inhaled AZD8871 600 μg in patients with moderate to severe COPD
Time Frame: Day 1 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | AZD8871 | Anoro® Ellipta® | Placebo
Number analyzed (Participants) | 70 | 69 | 68
Liters
  Day 1: number analyzed (Participants) | 69 | 68 | 68
  Day 1 | 0.3072 (0.1565) | 0.2798 (0.1695) | 0.0230 (0.0923)
  Day 14: number analyzed (Participants) | 70 | 67 | 67
  Day 14 | 0.3394 (0.2462) | 0.3102 (0.1998) | 0.0021 (0.1204)

4. Secondary Outcome: FEV1 AUC(0-12)/12h (Area Under the Curve for the Change in FEV1 From Baseline to 12h, Normalised by the Time Window)
Description: To evaluate the efficacy of inhaled AZD8871 600 μg in patients with moderate to severe COPD
Time Frame: Day 1 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | AZD8871 | Anoro® Ellipta® | Placebo
Number analyzed (Participants) | 70 | 69 | 68
Liters
  Day 1: number analyzed (Participants) | 69 | 69 | 68
  Day 1 | 0.2668 (0.1494) | 0.2720 (0.1697) | 0.0096 (0.0946)
  Day 14: number analyzed (Participants) | 69 | 68 | 67
  Day 14 | 0.3024 (0.2141) | 0.2919 (0.2027) | -0.0032 (0.1150)

5. Secondary Outcome: FEV1 AUC(0-24)/24h (Area Under the Curve for the Change in FEV1 From Baseline to 24h, Normalised by the Time Window)
Description: To evaluate the efficacy of inhaled AZD8871 600 μg in patients with moderate to severe COPD
Time Frame: Day 1 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | AZD8871 | Anoro® Ellipta® | Placebo
Number analyzed (Participants) | 70 | 69 | 68
Liters
  Day 1: number analyzed (Participants) | 69 | 69 | 68
  Day 1 | 0.1832 (0.1399) | 0.2333 (0.1742) | -0.0132 (0.0920)
  Day 14: number analyzed (Participants) | 70 | 68 | 67
  Day 14 | 0.2223 (0.2154) | 0.2417 (0.2012) | -0.0324 (0.1104)

6. Secondary Outcome: Change From Baseline in Trough FEV1 on Day 2 and Day 8.
Description: To evaluate the efficacy of inhaled AZD8871 600 μg in patients with moderate to severe COPD
Time Frame: Day 2 and Day 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | AZD8871 | Anoro® Ellipta® | Placebo
Number analyzed (Participants) | 70 | 69 | 68
Liters
  Day 2: number analyzed (Participants) | 69 | 69 | 68
  Day 2 | 0.1359 (0.1672) | 0.2249 (0.1897) | 0.0339 (0.1139)
  Day 8 | 0.2161 (0.1613) | 0.2748 (0.1894) | 0.0121 (0.1240)
Statistical Analysis 1: Comparison: AZD8871 vs Placebo; Day 2; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.098, 95% CI 2-sided [0.051 to 0.146]
Statistical Analysis 2: Comparison: AZD8871 vs Placebo; Day 8; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.195, 95% CI 2-sided [0.148 to 0.242]

7. Secondary Outcome: Change From Baseline in Peak FEV1 on Day 1, Day 8 and Day 14.
Description: To evaluate the efficacy of inhaled AZD8871 600 μg in patients with moderate to severe COPD
Time Frame: At Day 1, Day 8, and Day 14.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | AZD8871 | Anoro® Ellipta® | Placebo
Number analyzed (Participants) | 70 | 69 | 68
Liters
  Day 1: number analyzed (Participants) | 69 | 69 | 68
  Day 1 | 0.403 (0.182) | 0.333 (0.176) | 0.092 (0.086)
  Day 8 | 0.511 (0.240) | 0.454 (0.227) | 0.120 (0.130)
  Day 14: number analyzed (Participants) | 70 | 68 | 67
  Day 14 | 0.464 (0.255) | 0.391 (0.215) | 0.066 (0.131)
Statistical Analysis 1: Comparison: AZD8871 vs Placebo; Day 1; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.306, 95% CI 2-sided [0.266 to 0.346]
Statistical Analysis 2: Comparison: AZD8871 vs Placebo; Day 8; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.374, 95% CI 2-sided [0.324 to 0.425]
Statistical Analysis 3: Comparison: AZD8871 vs Placebo; Day 14; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.388, 95% CI 2-sided [0.329 to 0.447]

8. Secondary Outcome: Change From Baseline in Breathlessness, Cough and Sputum Scale (BCSS) Total Score at Day 1 to Day 8, Day 9 to Day 14, Day 1 to Day 14
Description: To evaluate the efficacy of inhaled AZD8871 600 μg in patients with moderate to severe COPD. The BCSS questionnaire is a 3-item, patient-reported outcome (PRO) measure. On a daily basis, patients are asked to evaluate each of their 3 symptoms (breathlessness, cough, and sputum) on a 5-point Likert scale ranging from 0 to 4, with higher scores indicating a higher severity of the symptom. The BCSS questionnaire is expressed as a daily total score, which is the sum of the 3 symptom scores, ranging from 0 to 12.
Time Frame: Day 1 to Day 8, Day 9 to Day 14, Day 1 to Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AZD8871 | Anoro® Ellipta® | Placebo
Number analyzed (Participants) | 70 | 69 | 68
Score on a scale
  Day 1 to Day 8: number analyzed (Participants) | 70 | 69 | 66
  Day 1 to Day 8 | -0.37 (1.27) | -0.61 (1.31) | 0.16 (1.11)
  Day 9 to Day 14 | -0.35 (1.58) | -0.63 (1.49) | 0.53 (1.43)
  Day 1 to Day 14 | -0.36 (1.33) | -0.63 (1.32) | 0.36 (1.26)
Statistical Analysis 1: Comparison: AZD8871 vs Placebo; Day 1 to Day 8; Test type: Superiority; p = 0.0010, Mixed Models Analysis; Mean Difference (Final Values) = -0.551, 95% CI 2-sided [-0.876 to -0.226]
Statistical Analysis 2: Comparison: AZD8871 vs Placebo; Day 9 to Day 14; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.867, 95% CI 2-sided [-1.248 to -0.486]
Statistical Analysis 3: Comparison: AZD8871 vs Placebo; Day 1 to Day 14; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.722, 95% CI 2-sided [-1.047 to -0.397]

9. Primary Outcome: Change From Baseline in Chronic Obstructive Pulmonary Disease (COPD) Assessment Test (CAT) at Day 1 to Day 8, Day 9 to Day 14, Day 1 to Day 14
Description: To evaluate the efficacy of inhaled AZD8871 600 μg in patients with moderate to severe COPD. At each visit, patients are asked to evaluate the impact of COPD on their wellbeing and daily life on a 6-point Likert scale ranging from 0 to 5, with higher scores indicating a higher impact of COPD. The CAT is expressed as a total score, which is a sum of the 8 questions, ranging from 0 to 40.
Time Frame: Day 1 to Day 8, Day 9 to Day 14, Day 1 to Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AZD8871 | Anoro® Ellipta® | Placebo
Number analyzed (Participants) | 70 | 69 | 68
Score on a scale
  Day 1 to Day 8: number analyzed (Participants) | 68 | 65 | 65
  Day 1 to Day 8 | -2.11 (4.34) | -2.78 (4.34) | -0.57 (4.69)
  Day 9 to Day 14: number analyzed (Participants) | 68 | 65 | 67
  Day 9 to Day 14 | -2.87 (5.01) | -3.29 (4.94) | -0.52 (5.06)
  Day 1 to Day 14: number analyzed (Participants) | 68 | 65 | 67
  Day 1 to Day 14 | -2.42 (4.49) | -3.01 (4.51) | -0.59 (4.81)
Statistical Analysis 1: Comparison: AZD8871 vs Placebo; Day 1 to Day 8; Test type: Superiority; p = 0.0022, Mixed Models Analysis; Mean Difference (Final Values) = -1.571, 95% CI 2-sided [-2.563 to -0.579]
Statistical Analysis 2: Comparison: AZD8871 vs Placebo; Day 9 to Day 14; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.386, 95% CI 2-sided [-3.541 to -1.230]
Statistical Analysis 3: Comparison: AZD8871 vs Placebo; Day 1 to Day 14; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = -1.912, 95% CI 2-sided [-2.923 to -0.901]

10. Secondary Outcome: Number of Participants With Adverse Events.
Description: To evaluate the safety and tolerability of inhaled AZD8871 600 μg in patients with moderate to severe COPD
Time Frame: From Screening to folow-up or discontinuation (42 days after last study drug)
Measure: Number; unit: Participants
Arm/Group | AZD8871 | Anoro® Ellipta® | Placebo
Number analyzed (Participants) | 70 | 69 | 68
Participants
  Any AE | 39 | 38 | 35
  Any AE with outcome=death | 0 | 0 | 0
  Any SAE (including events with outcome=death) | 0 | 2 | 2
  Any AE leading to discontinuation of treatment | 0 | 1 | 0
  Any AE leading to withdrawal from study | 0 | 1 | 0

11. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: To investigate the Cmax of AZD8871 600 μg and its primary metabolite after multiple dose administration of inhaled AZD8871 in patients with moderate to severe COPD
Time Frame: At Day 1 and Day 14 (at pre-dose and at 30 minutes (min), 1, 2, 4, 6, 8, 12, and 24 hours post-dose)
Population: PK analysis set (PKS): All participants participating in the subset of the PK participants, who received at least 1 dose of AZD8871 600 μg.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | AZD8871
Number analyzed (Participants) | 70
pg/mL
  AZD8871 - Day 1: number analyzed (Participants) | 41
  AZD8871 - Day 1 | 310.4 (61.30)
  AZD8871 - Day 14: number analyzed (Participants) | 41
  AZD8871 - Day 14 | 532.9 (46.58)
  LAS191861- Day 1: number analyzed (Participants) | 41
  LAS191861- Day 1 | 26.64 (53.33)
  LAS191861- Day 14: number analyzed (Participants) | 41
  LAS191861- Day 14 | 63.29 (52.12)

12. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Description: To investigate the Tmax of AZD8871 600 μg and its primary metabolite after multiple dose administration of inhaled AZD8871 in patients with moderate to severe COPD
Time Frame: At Day 1 and Day 14 (at pre-dose and at 30 minutes (min), 1, 2, 4, 6, 8, 12, and 24 hours post-dose)
Population: as for outcome 11
Measure: Median (Full Range); unit: Hours
Arm/Group | AZD8871
Number analyzed (Participants) | 70
Hours
  AZD8871- Day 1: number analyzed (Participants) | 41
  AZD8871- Day 1 | 0.99 [0.38 to 2.02]
  AZD8871- Day 14: number analyzed (Participants) | 41
  AZD8871- Day 14 | 0.98 [0.45 to 2.05]
  LAS191861 - Day 1: number analyzed (Participants) | 41
  LAS191861 - Day 1 | 2.00 [0.98 to 4.00]
  LAS191861 - Day 14: number analyzed (Participants) | 41
  LAS191861 - Day 14 | 2.00 [0.98 to 4.03]

13. Secondary Outcome: Time to Reach Last Quantifiable Plasma Concentration (Tlast)
Description: To investigate the Tlast of AZD8871 600 μg and its primary metabolite after multiple dose administration of inhaled AZD8871 in patients with moderate to severe COPD
Time Frame: At Day 1 and Day 14 (at pre-dose and at 30 minutes (min), 1, 2, 4, 6, 8, 12, and 24 hours post-dose)
Population: as for outcome 11
Measure: Median (Full Range); unit: Hours
Arm/Group | AZD8871
Number analyzed (Participants) | 70
Hours
  AZD8871 -Day 1: number analyzed (Participants) | 41
  AZD8871 -Day 1 | 23.93 [7.98 to 24.05]
  AZD8871-Day 14: number analyzed (Participants) | 41
  AZD8871-Day 14 | 24.03 [23.90 to 24.37]
  LAS191861 - Day 1: number analyzed (Participants) | 41
  LAS191861 - Day 1 | 23.92 [1.97 to 24.05]
  LAS191861 - Day 14: number analyzed (Participants) | 41
  LAS191861 - Day 14 | 24.03 [23.90 to 24.37]

14. Secondary Outcome: Area Under the Plasma Concentration-curve From Time 0 to the Time of Last Quantifiable Concentration (AUClast)
Description: To investigate the AUClast of AZD8871 600 μg and its primary metabolite after multiple dose administration of inhaled AZD8871 in patients with moderate to severe COPD
Time Frame: At Day 1 and Day 14 (at pre-dose and at 30 minutes (min), 1, 2, 4, 6, 8, 12, and 24 hours post-dose)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | AZD8871
Number analyzed (Participants) | 70
h*pg/mL
  AZD8871- Day 1: number analyzed (Participants) | 41
  AZD8871- Day 1 | 1655 (85.24)
  AZD8871-Day 14: number analyzed (Participants) | 41
  AZD8871-Day 14 | 4001 (55.64)
  LAS191861 -Day 1: number analyzed (Participants) | 41
  LAS191861 -Day 1 | 251.9 (97.81)
  LAS191861 -Day 14: number analyzed (Participants) | 41
  LAS191861 -Day 14 | 943.3 (63.08)

15. Secondary Outcome: Area Under the Plasma Concentration-curve From Time 0 to 24 Hours Post-dose [AUC(0-24)]
Description: To investigate the AUC(0-24) of AZD8871 600 μg and its primary metabolite after multiple dose administration of inhaled AZD8871 in patients with moderate to severe COPD
Time Frame: At Day 1 and Day 14 (at pre-dose and at 30 minutes (min), 1, 2, 4, 6, 8, 12, and 24 hours post-dose)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | AZD8871
Number analyzed (Participants) | 70
h*pg/mL
  AZD8871- Day 1: number analyzed (Participants) | 41
  AZD8871- Day 1 | 1661 (83.55)
  AZD8871- Day 14: number analyzed (Participants) | 41
  AZD8871- Day 14 | 3996 (55.66)
  LAS191861 - Day 1: number analyzed (Participants) | 41
  LAS191861 - Day 1 | 289.5 (57.83)
  LAS191861 - Day 14: number analyzed (Participants) | 41
  LAS191861 - Day 14 | 941.7 (63.11)

16. Secondary Outcome: Average Plasma Concentration During a Dosing Interval (Cavg)
Description: To investigate the Cavg of AZD8871 600 μg and its primary metabolite after multiple dose administration of inhaled AZD8871 in patients with moderate to severe COPD
Time Frame: At Day 14 (at pre-dose and at 30 minutes (min), 1, 2, 4, 6, 8, 12, and 24 hours post-dose)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | AZD8871
Number analyzed (Participants) | 70
pg/mL
  AZD8871 -Day 14: number analyzed (Participants) | 41
  AZD8871 -Day 14 | 166.5 (55.63)
  LAS191861 - Day 14: number analyzed (Participants) | 41
  LAS191861 - Day 14 | 39.23 (63.06)

17. Secondary Outcome: Fluctuation Index During a Dosing Interval (%Fluctuation)
Description: To investigate the %Fluctuation of AZD8871 600 μg and its primary metabolite after multiple dose administration of inhaled AZD8871 in patients with moderate to severe COPD. Fluctuation index during a dosing interval is estimated as 100*(Cmax - Cmin)/Cavg (%), where Cmin is the minimum concentration at the end of the dosing interval.
Time Frame: At Day 14 (at pre-dose and at 30 minutes (min), 1, 2, 4, 6, 8, 12, and 24 hours post-dose)
Population: as for outcome 11
Measure: Median (Full Range); unit: percentage of fluctuation
Arm/Group | AZD8871
Number analyzed (Participants) | 70
percentage of fluctuation
  AZD8871- Day 14: number analyzed (Participants) | 41
  AZD8871- Day 14 | 273.1 [128 to 514]
  LAS191861 - Day 14: number analyzed (Participants) | 41
  LAS191861 - Day 14 | 91.03 [39.3 to 174]

18. Secondary Outcome: Accumulation Ratio for Cmax (Rac(Cmax))
Description: To investigate the Rac (Cmax) of AZD8871 600 μg and its primary metabolite after multiple dose administration of inhaled AZD8871 in patients with moderate to severe COPD. Accumulation ratio for Cmax estimated as (Cmax on Day 14/Cmax on Day 1).
Time Frame: At Day 14
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | AZD8871
Number analyzed (Participants) | 70
Ratio
  AZD8871 -Day 14: number analyzed (Participants) | 41
  AZD8871 -Day 14 | 1.725 (44.77)
  LAS191861 - Day 14: number analyzed (Participants) | 41
  LAS191861 - Day 14 | 2.377 (40.02)

19. Secondary Outcome: Accumulation Ratio for AUC(0-24) Rac(AUC(0-24))
Description: To investigate the Rac(AUC(0-24) of AZD8871 600 μg and its primary metabolite after multiple dose administration of inhaled AZD8871 in patients with moderate to severe COPD. Accumulation ratio for AUC0-24 estimated as (AUC0-24 on Day 14/AUC0-24 on Day 1).
Time Frame: At Day 14
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | AZD8871
Number analyzed (Participants) | 70
Ratio
  AZD8871 - Day 14: number analyzed (Participants) | 41
  AZD8871 - Day 14 | 2.406 (50.37)
  LAS191861 -Day 14: number analyzed (Participants) | 41
  LAS191861 -Day 14 | 3.443 (47.15)

20. Secondary Outcome: Change From Baseline in Use of Rescue Medication
Description: To evaluate the efficacy of inhaled AZD8871 600 μg in patients with moderate to severe COPD
Time Frame: Day 1 to Day 8 and Day 9 to Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of use
Arm/Group | AZD8871 | Anoro® Ellipta® | Placebo
Number analyzed (Participants) | 70 | 69 | 68
Percentage of use
  Day 1 to Day 8: number analyzed (Participants) | 69 | 65 | 64
  Day 1 to Day 8 | -1.00 (1.83) | -0.95 (2.03) | 0.18 (2.13)
  Day 9 to Day 14: number analyzed (Participants) | 70 | 67 | 68
  Day 9 to Day 14 | -0.78 (1.97) | -0.87 (1.96) | 0.52 (1.80)
Statistical Analysis 1: Comparison: AZD8871 vs Placebo; Day 1 to Day 8; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.268, 95% CI 2-sided [-1.741 to -0.794]
Statistical Analysis 2: Comparison: AZD8871 vs Placebo; Day 9 to Day 14; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.302, 95% CI 2-sided [-1.804 to -0.800]

ADVERSE EVENTS:
Time Frame: AEs starting on or after the first administration of study treatment, up to and including 42 days after the last dose of study treatment.
Description: An adverse event was the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition might be symptoms, signs or the abnormal results of an investigation. The safety population was defined as all randomized patients who took at least one dose of IMP.
Arm/Group | AZD8871 | Anoro® Ellipta® | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/69 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/70 | 2/69 | 2/68
Other Adverse Events (participants affected / at risk) | 19/70 | 19/69 | 17/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD8871 (N=70) | Anoro® Ellipta® (N=69) | Placebo (N=68)
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD8871 (N=70) | Anoro® Ellipta® (N=69) | Placebo (N=68)
Headache (Nervous system disorders) | 14 | 13 | 14
Nasopharyngitis (Infections and infestations) | 6 | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT03645434/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT03645434/SAP_001.pdf